CLINICAL TRIAL: NCT00039858
Title: Evaluation of Argatroban Injection in Pediatric Patients Requiring Anticoagulant Alternatives to Heparin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Encysive Pharmaceuticals (Industry)
Collaborators: GlaxoSmithKline (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARG-401; SKF105043/013
Record Dates: First submitted 2002-06-13; First posted 2002-06-14 (Estimated); Last update posted 2007-01-11 (Estimated); Status verified 2007-01

CONDITIONS: Thrombocytopenia; Thrombosis
Keywords: heparin-induced thrombocytopenia; heparin-induced thrombocytopenia and thrombosis; HIT; HITTS; anticoagulation
MeSH Terms: conditions — Thrombocytopenia; Thrombosis | interventions — argatroban

INTERVENTIONS:
Drug: Argatroban

SUMMARY:
The purpose of this study is to evaluate the safe and effective dose of Argatroban for prophylaxis and/or treatment of thrombosis in pediatric patients with current or previous diagnosis of heparin-induced thrombocytopenia (HIT) and thrombosis syndrome (HITTS), or who in the opinion of the investigator require alternative anticoagulation due to an underlying condition.

ELIGIBILITY:
Criteria for Inclusion:

* Males and females ages birth to 16 years,inclusive, at enrollment. For neonates, the minimum corrected gestational age should be 37 weeks.
* Documented HIT defined as a fall in platelet count to less than 100,000/uL or a >=50% decrease in platelets after the initiation of heparin therapy with no apparent explanation other than HIT, or
* Require anticoagulation and have a documented history of a positive HIT test in the absence of current thrombocytopenia (i.e. patients at risk for HIT), or
* In the opinion of the investigator, require alternative anticoagulation due to an underlying condition, such as AT-III deficiency or heparin resistance.
* Signed (written) informed consent or assent by the patient (if age appropriate) and the patient's parent or guardian.

Criteria for Exclusion:

* Any condition which, in the investigator's opinion, would contraindicate the use of Argatroban or would endanger the patient if he/she participated in this trial.
* Unexplained aPTT > 2 times the upper limit of normal at baseline, in the absence of heparin.
* International Normalized Ratio (INR) >1.6 at baseline in the absence of warfarin.
* Known clinical site of bleeding or predisposition to bleeding (e.g., GI bleed, hematuria, hemorrhagic CVA,retroperitoneal hematoma, diabetic retinopathy, hemorrhagic pericardial effusion, or hemorrhagic pleural effusion. Patients who have a known clinical site of bleeding may be enrolled if the investigator deems the risk of continued thrombosis to outweigh the potential bleeding risk.
* Any patient who has received any investigational medication within 30 days prior to the first dose of study medication or who is scheduled to receive an investigational drug other than Argatroban during the course of the study.
* Known hypersensitivity to Argatroban or chemically related compounds.
* Females of childbearing potential who are pregnant (positive serum beta-HCG), breast feeding, or sexually active and not taking adequate contraceptive precautions (e.g. IUD or oral contraceptives).
* Any patient receiving a thrombolytic medication (e.g. tPA).
* Any neonate with a corrected gestational age of < or = 44 weeks and bleeding in the head (Grade I or above) as determined by head ultrasound.

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24
Dates: Start 2003-09; Study Completion 2006-03

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Mattel Children's Hospital at UCLA, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago Children's Hospital, Chicago, Illinois
  - Children's Hospital of Illinois, Peoria, Illinois
  - Kosair Children's Hospital, University of Louisville, Louisville, Kentucky
  - Children's Hospital of Boston, Boston, Massachusetts
  - Michigan Congenital Heart Center, Ann Arbor, Michigan
  - Rainbow Babies at Children's Hospital, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Children's Hospital and Regional Medical Center, Seattle, Washington